CLINICAL TRIAL: NCT00659698
Title: Prevention for Surgical Site Infection After Hepatic Resection
Brief Title: Effect of an Artificial Pancreas in Patients Undergoing Hepatic Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Kochi University, Kochi Medical School
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TGC-AP-02; Kochi University
Record Dates: First submitted 2008-04-11; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Liver Diseases
Keywords: surgical; site; infection
MeSH Terms: conditions — Liver Diseases; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): received programmed infusions of insulin determined by the control algorithm of the artificial pancreas
  Interventions: Device: the closed-loop STG-22 system (Nikkiso Inc, Tokyo, Japan)
- 2 (No Intervention): glucose levels were controlled using a manual injection of insulin according to the commonly used sliding scale

INTERVENTIONS:
Device: the closed-loop STG-22 system (Nikkiso Inc, Tokyo, Japan) — artificial pancreas
  Other Names: an artificial pancreas system (Nikkiso Inc, Tokyo, Japan)
  Arms: 1

SUMMARY:
This study evaluated that strict control of perioperative blood glucose following hepatic resection by using an artificial pancreas would improve postoperative surgical site infection.

DETAILED DESCRIPTION:
This study recruited 70 patients undergoing elective hepatic resection for liver diseases. Perioperative blood glucose concentration was continuously monitored using an artificial pancreas system. We prospectively divided patients into two groups: one for whom glucose levels were controlled using a manual injection of insulin according to the commonly used sliding scale and another that received programmed infusions of insulin determined by the control algorithm of the artificial pancreas.

ELIGIBILITY:
Inclusion Criteria:

* This study recruited 70 patients undergoing elective hepatic resection for liver diseases. Perioperative blood glucose concentration was continuously monitored using an artificial pancreas system.

Exclusion Criteria:

* weight loss greater than 10% during the previous 6 months, signs of distant metastasis, and respiratory, renal, or heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
the incidence of surgical site infection | 30th postoperative day

SECONDARY OUTCOMES:
the incidence of hypoglycemia and cost during the hospitalization | during the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Takehiro Okabayashi, MD, Study Director — Kochi Medical School
Locations (1):
- Kochi Medical School, Nankoku, Kochi, Japan